CLINICAL TRIAL: NCT03615131
Title: Accuracy of Multi-parametric Prostate MRI and MRI-targeted, Ultrasound-navigated Prostate Fusion Biopsy in the Detection of Prostate Cancer:
Brief Title: Accuracy of mpMRI and MRI-targeted, Ultrasound-navigated Prostate Fusion Biopsy in Detection of Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01098
Record Dates: First submitted 2018-07-16; First posted 2018-08-03 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; mpMRI-TRUS fusion biopsy; PIRADS; Gleason score
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Prostate biopsies without DNA evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI-TRUS fusion prostate biopsy: Single Arm Study, MRI and Prostate-Biopsy on same patient, individual patient acts as own control for intervention
  Interventions: Diagnostic Test: MRI-TRUS fusion prostate biopsy

INTERVENTIONS:
Diagnostic Test: MRI-TRUS fusion prostate biopsy — First an advanced MRI prostate image is obtained, annotated and recorded by the Radiology of the Kantonsspital Winterthur. Next, using special fusion technology, the recorded MRI image is fused with a live transrectal ultrasound by the Urologist who performs a MRI/TRUS fusion biopsy.
  Other Names: MRI prior to biopsy

SUMMARY:
The investigators examined whether a high PI-RADS v2 score correlates with the presence of prostate cancer. In addition, the investigator inspected whether the lesion size as determined by mpMRI correlates with the presence of prostate cancer. Furthermore, the investigators study aimed to determine the sensitivity and specificity of mpMRI with respect to prostate carcinoma detection.

DETAILED DESCRIPTION:
Purpose: In recent years, multiparametric Magnet Resonance Imaging (mpMRI) has been established as a diagnostic imaging technique of the prostate and its assessment standardized with the "prostate imaging - data and reporting system" (PI-RADS v2). The previously established Likert scale from 1 to 5 has been shown to reflect the increasing probability of a carcinoma. Suspicious MRI lesions can be biopsied in a targeted fashion using ultrasound navigation termed fusion biopsy. The investigators examined whether a high PI-RADS v2 score correlates with the presence of prostate cancer. In addition, the investigators inspected whether the lesion size as determined by mpMRI correlates with the presence of prostate cancer. Furthermore, the investigators study aimed to determine the sensitivity and specificity of mpMRI with respect to prostate carcinoma detection.

Materials and Methods: This prospective study includes 228 consecutive patients, which underwent a perineal MRI-TRUS-fused prostate biopsy (BiopSee®, MedCom Company) during the period of September 2015 to March 2017 at the cantonal hospital Winterthur due to a suspicious PSA value, a suspicious digital rectal examination or a known prostate cancer under active surveillance. 71 patients were excluded due to lack of PI-RADS v2 diagnosis and / or MRI performed at a different center. Targeted biopsies were performed specifically in the indicated MRI lesions and standardized over the rest of the prostate (system biopsy).

ELIGIBILITY:
Inclusion Criteria:

* Patients with mRI-TRUS Fusion prostate biopsy
* age > 18y
* elevated PSA
* suspicious DRE (digital rectal examination)
* patients with prostate cancer under active surveillance

Exclusion Criteria:

* age < 18y
* treated prostate cancer (Radiotherapy, antiandrogens therapy, brachytherapy, HIFU).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men with a suspicious prostate cancer screening for the early detection of prostate cancer (PSA> 4 ng / ml, PSA velocity> 0.75 ng / ml / y or pathological DRE) or a planned re-biopsy in the context of active surveillance with known very-low-risk prostate cancer.
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Gleason score (minimum 2 to maximum of 10) | 01.09.2015 - 30.03.2017
  Histological grade of the glandular structures of prostate cancer tissue or the difference in appearance compared with a normal structure.
  Pattern 1 - corresponds to a well differentiated carcinoma. Pattern 2 - corresponds to a moderately differentiated carcinoma. Pattern 3 - invade the surrounding tissue or having an infiltrative pattern; corresponds to a moderately differentiated carcinoma.
  Pattern 4 - corresponds to a poorly differentiated carcinoma. Pattern 5 - corresponds to an anaplastic carcinoma.
  The pathologist then sums the pattern-number of the primary and secondary grades to obtain the final Gleason score.
  Gleason scores range from 2 to 10, with 2 representing the most well-differentiated tumors and 10 the least-differentiated tumors.
ISUP (International Society of Urological Pathology) Grading Group (Grade 1 to Grade 5) | 01.09.2015 - 30.03.2017
  New grading system for histological grade of the glandular structures of prostate cancer tissue or the difference in appearance compared with a normal structure
  Grade Group 1 (Gleason score ≤6) - Only individual discrete well-formed glands Grade Group 2 (Gleason score 3+4=7) - Predominantly well-formed glands with a lesser component of poorly-formed/fused/cribriform glands Grade Group 3 (Gleason score 4+3=7) - Predominantly poorly-formed/fused/cribriform glands with a lesser component of well-formed glands Grade Group 4 (Gleason score 8)
  * Only poorly-formed/fused/cribriform glands or
  * Predominantly well-formed glands with a lesser component lacking glands or
  * Predominantly lacking glands with a lesser component of well-formed glands Grade Group 5 (Gleason scores 9-10) - Lacks gland formation (or with necrosis) with or without poorly-formed/fused/cribriform glands
lesion volume (ml) | 01.09.2015 - 30.03.2017
  millilitre; size of suspected areas in prostate gland in MRI
PI-RADS v2 (Prostate Imaging Reporting and Data System Version 2) score (1 - 5) | 01.09.2015 - 30.03.2017
  Radiological grading system of prostate lesions in mpMRI
  The PI-RADS v2 system is designed to standardize image acquisition and reporting, and to be used by medical professionals in the initial evaluation of patients to assess the risk of clinically significant prostate cancer that may require biopsy and treatment.
  The scale is based on a score "Yes" or "No" for Dynamic Contrast-Enhanced (DCE) parameter, and from 1 to 5 for T2-weighted (T2W) and Diffusion-weighted imaging (DWI). The score is given for each lesion, with 1 being most probably benign and 5 being highly suspicious of malignancy:
  PI-RADS 1: very low (clinically significant cancer is highly unlikely to be present) PI-RADS 2: low (clinically significant cancer is unlikely to be present) PI-RADS 3: intermediate (clinically significant cancer is equivocal) PI-RADS 4: high (clinically significant cancer is likely to be present) PI-RADS 5: very high (clinically significant cancer is highly likely to be present)
Prostate specific antigen (PSA) | 01.09.2015 - 30.03.2017
  ng per ml; enzyme secreted by the prostate gland
Digital rectal examination (DRE) | 01.09.2015 - 30.03.2017
  consistence of prostate gland
Prostate specific antigen - density | 01.09.2015 - 30.03.2017
  ng per ml per ml; The relationship of the prostate specific antigen level to the size and weight (volume) of the prostate.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Urologie Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel R, DeSantis C, Virgo K, Stein K, Mariotto A, Smith T, Cooper D, Gansler T, Lerro C, Fedewa S, Lin C, Leach C, Cannady RS, Cho H, Scoppa S, Hachey M, Kirch R, Jemal A, Ward E. Cancer treatment and survivorship statistics, 2012. CA Cancer J Clin. 2012 Jul-Aug;62(4):220-41. doi: 10.3322/caac.21149. Epub 2012 Jun 14. PMID 22700443
- [Background] Heidenreich A, Bastian PJ, Bellmunt J, Bolla M, Joniau S, van der Kwast T, Mason M, Matveev V, Wiegel T, Zattoni F, Mottet N; European Association of Urology. EAU guidelines on prostate cancer. part 1: screening, diagnosis, and local treatment with curative intent-update 2013. Eur Urol. 2014 Jan;65(1):124-37. doi: 10.1016/j.eururo.2013.09.046. Epub 2013 Oct 6. PMID 24207135
- [Background] Hoeks CM, Barentsz JO, Hambrock T, Yakar D, Somford DM, Heijmink SW, Scheenen TW, Vos PC, Huisman H, van Oort IM, Witjes JA, Heerschap A, Futterer JJ. Prostate cancer: multiparametric MR imaging for detection, localization, and staging. Radiology. 2011 Oct;261(1):46-66. doi: 10.1148/radiol.11091822. PMID 21931141
- [Background] Hamoen EHJ, de Rooij M, Witjes JA, Barentsz JO, Rovers MM. Use of the Prostate Imaging Reporting and Data System (PI-RADS) for Prostate Cancer Detection with Multiparametric Magnetic Resonance Imaging: A Diagnostic Meta-analysis. Eur Urol. 2015 Jun;67(6):1112-1121. doi: 10.1016/j.eururo.2014.10.033. Epub 2014 Nov 6. PMID 25466942
- [Background] Weinreb JC, Barentsz JO, Choyke PL, Cornud F, Haider MA, Macura KJ, Margolis D, Schnall MD, Shtern F, Tempany CM, Thoeny HC, Verma S. PI-RADS Prostate Imaging - Reporting and Data System: 2015, Version 2. Eur Urol. 2016 Jan;69(1):16-40. doi: 10.1016/j.eururo.2015.08.052. Epub 2015 Oct 1. PMID 26427566
- [Background] Barentsz JO, Richenberg J, Clements R, Choyke P, Verma S, Villeirs G, Rouviere O, Logager V, Futterer JJ; European Society of Urogenital Radiology. ESUR prostate MR guidelines 2012. Eur Radiol. 2012 Apr;22(4):746-57. doi: 10.1007/s00330-011-2377-y. Epub 2012 Feb 10. PMID 22322308
- [Background] Renard Penna R, Brenot-Rossi I, Salomon L, Soulie M. [Prostate cancer imaging: MRI and nuclear imaging]. Prog Urol. 2015 Nov;25(15):933-46. doi: 10.1016/j.purol.2015.07.016. French. PMID 26519961
- [Background] Roethke MC, Kuru TH, Schultze S, Tichy D, Kopp-Schneider A, Fenchel M, Schlemmer HP, Hadaschik BA. Evaluation of the ESUR PI-RADS scoring system for multiparametric MRI of the prostate with targeted MR/TRUS fusion-guided biopsy at 3.0 Tesla. Eur Radiol. 2014 Feb;24(2):344-52. doi: 10.1007/s00330-013-3017-5. Epub 2013 Oct 3. PMID 24196383
- [Background] Schimmoller L, Quentin M, Arsov C, Lanzman RS, Hiester A, Rabenalt R, Antoch G, Albers P, Blondin D. Inter-reader agreement of the ESUR score for prostate MRI using in-bore MRI-guided biopsies as the reference standard. Eur Radiol. 2013 Nov;23(11):3185-90. doi: 10.1007/s00330-013-2922-y. Epub 2013 Jun 12. PMID 23756958
- [Background] Kuru TH, Herden J, Zugor V, Akbarov I, Pfister D, Porres D, Heidenreich A. How to Perform Image-guided Prostate Biopsy: In-bore and Fusion Approaches. Eur Urol Focus. 2016 Jun;2(2):151-153. doi: 10.1016/j.euf.2016.03.016. Epub 2016 Apr 12. PMID 28723529
- [Background] Arsov C, Rabenalt R, Blondin D, Quentin M, Hiester A, Godehardt E, Gabbert HE, Becker N, Antoch G, Albers P, Schimmoller L. Prospective randomized trial comparing magnetic resonance imaging (MRI)-guided in-bore biopsy to MRI-ultrasound fusion and transrectal ultrasound-guided prostate biopsy in patients with prior negative biopsies. Eur Urol. 2015 Oct;68(4):713-20. doi: 10.1016/j.eururo.2015.06.008. Epub 2015 Jun 23. PMID 26116294
- [Background] Quentin M, Blondin D, Arsov C, Schimmoller L, Hiester A, Godehardt E, Albers P, Antoch G, Rabenalt R. Prospective evaluation of magnetic resonance imaging guided in-bore prostate biopsy versus systematic transrectal ultrasound guided prostate biopsy in biopsy naive men with elevated prostate specific antigen. J Urol. 2014 Nov;192(5):1374-9. doi: 10.1016/j.juro.2014.05.090. Epub 2014 May 24. PMID 24866597
- [Background] Vargas HA, Hotker AM, Goldman DA, Moskowitz CS, Gondo T, Matsumoto K, Ehdaie B, Woo S, Fine SW, Reuter VE, Sala E, Hricak H. Updated prostate imaging reporting and data system (PIRADS v2) recommendations for the detection of clinically significant prostate cancer using multiparametric MRI: critical evaluation using whole-mount pathology as standard of reference. Eur Radiol. 2016 Jun;26(6):1606-12. doi: 10.1007/s00330-015-4015-6. Epub 2015 Sep 22. PMID 26396111
- [Background] Samaratunga H, Delahunt B, Yaxley J, Srigley JR, Egevad L. From Gleason to International Society of Urological Pathology (ISUP) grading of prostate cancer. Scand J Urol. 2016 Oct;50(5):325-9. doi: 10.1080/21681805.2016.1201858. Epub 2016 Jul 14. PMID 27415753
- [Background] Egevad L, Delahunt B, Srigley JR, Samaratunga H. International Society of Urological Pathology (ISUP) grading of prostate cancer - An ISUP consensus on contemporary grading. APMIS. 2016 Jun;124(6):433-5. doi: 10.1111/apm.12533. PMID 27150257
- [Background] Epstein JI, Egevad L, Amin MB, Delahunt B, Srigley JR, Humphrey PA; Grading Committee. The 2014 International Society of Urological Pathology (ISUP) Consensus Conference on Gleason Grading of Prostatic Carcinoma: Definition of Grading Patterns and Proposal for a New Grading System. Am J Surg Pathol. 2016 Feb;40(2):244-52. doi: 10.1097/PAS.0000000000000530. PMID 26492179
- [Background] Martorana E, Pirola GM, Scialpi M, Micali S, Iseppi A, Bonetti LR, Kaleci S, Torricelli P, Bianchi G. Lesion volume predicts prostate cancer risk and aggressiveness: validation of its value alone and matched with prostate imaging reporting and data system score. BJU Int. 2017 Jul;120(1):92-103. doi: 10.1111/bju.13649. Epub 2016 Oct 4. PMID 27608292
- [Background] Le JD, Tan N, Shkolyar E, Lu DY, Kwan L, Marks LS, Huang J, Margolis DJ, Raman SS, Reiter RE. Multifocality and prostate cancer detection by multiparametric magnetic resonance imaging: correlation with whole-mount histopathology. Eur Urol. 2015 Mar;67(3):569-76. doi: 10.1016/j.eururo.2014.08.079. Epub 2014 Sep 23. PMID 25257029
- [Background] Schoots IG, Roobol MJ, Nieboer D, Bangma CH, Steyerberg EW, Hunink MG. Magnetic resonance imaging-targeted biopsy may enhance the diagnostic accuracy of significant prostate cancer detection compared to standard transrectal ultrasound-guided biopsy: a systematic review and meta-analysis. Eur Urol. 2015 Sep;68(3):438-50. doi: 10.1016/j.eururo.2014.11.037. Epub 2014 Dec 3. PMID 25480312
- [Background] Valerio M, Donaldson I, Emberton M, Ehdaie B, Hadaschik BA, Marks LS, Mozer P, Rastinehad AR, Ahmed HU. Detection of Clinically Significant Prostate Cancer Using Magnetic Resonance Imaging-Ultrasound Fusion Targeted Biopsy: A Systematic Review. Eur Urol. 2015 Jul;68(1):8-19. doi: 10.1016/j.eururo.2014.10.026. Epub 2014 Nov 1. PMID 25454618
- [Background] Siddiqui MM, Rais-Bahrami S, Truong H, Stamatakis L, Vourganti S, Nix J, Hoang AN, Walton-Diaz A, Shuch B, Weintraub M, Kruecker J, Amalou H, Turkbey B, Merino MJ, Choyke PL, Wood BJ, Pinto PA. Magnetic resonance imaging/ultrasound-fusion biopsy significantly upgrades prostate cancer versus systematic 12-core transrectal ultrasound biopsy. Eur Urol. 2013 Nov;64(5):713-719. doi: 10.1016/j.eururo.2013.05.059. Epub 2013 Jun 12. PMID 23787357
- [Background] Tewes S, Hueper K, Hartung D, Imkamp F, Herrmann TR, Weidemann J, Renckly S, Kuczyk MA, Wacker F, Peters I. Targeted MRI/TRUS fusion-guided biopsy in men with previous prostate biopsies using a novel registration software and multiparametric MRI PI-RADS scores: first results. World J Urol. 2015 Nov;33(11):1707-14. doi: 10.1007/s00345-015-1525-4. Epub 2015 Mar 14. PMID 25774003
- [Background] Zhang L, Tang M, Chen S, Lei X, Zhang X, Huan Y. A meta-analysis of use of Prostate Imaging Reporting and Data System Version 2 (PI-RADS V2) with multiparametric MR imaging for the detection of prostate cancer. Eur Radiol. 2017 Dec;27(12):5204-5214. doi: 10.1007/s00330-017-4843-7. Epub 2017 Jun 27. PMID 28656462
- [Background] Cash H, Maxeiner A, Stephan C, Fischer T, Durmus T, Holzmann J, Asbach P, Haas M, Hinz S, Neymeyer J, Miller K, Gunzel K, Kempkensteffen C. The detection of significant prostate cancer is correlated with the Prostate Imaging Reporting and Data System (PI-RADS) in MRI/transrectal ultrasound fusion biopsy. World J Urol. 2016 Apr;34(4):525-32. doi: 10.1007/s00345-015-1671-8. Epub 2015 Aug 21. PMID 26293117
- [Background] Liddell H, Jyoti R, Haxhimolla HZ. mp-MRI Prostate Characterised PIRADS 3 Lesions are Associated with a Low Risk of Clinically Significant Prostate Cancer - A Retrospective Review of 92 Biopsied PIRADS 3 Lesions. Curr Urol. 2015 Jul;8(2):96-100. doi: 10.1159/000365697. Epub 2015 Jul 10. PMID 26889125
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Martorana E, Micali S, Ghaith A, Reggiani Bonetti L, Sighinolfi MC, Galli R, Paterlini M, Bianchi G. Advantages of single-puncture transperineal saturation biopsy of prostate: analysis of outcomes in 125 patients using our scheme. Int Urol Nephrol. 2015 May;47(5):735-41. doi: 10.1007/s11255-015-0967-3. Epub 2015 Apr 8. PMID 25852022
- [Background] Sonn GA, Chang E, Natarajan S, Margolis DJ, Macairan M, Lieu P, Huang J, Dorey FJ, Reiter RE, Marks LS. Value of targeted prostate biopsy using magnetic resonance-ultrasound fusion in men with prior negative biopsy and elevated prostate-specific antigen. Eur Urol. 2014 Apr;65(4):809-15. doi: 10.1016/j.eururo.2013.03.025. Epub 2013 Mar 17. PMID 23523537
- [Background] Miyagawa T, Ishikawa S, Kimura T, Suetomi T, Tsutsumi M, Irie T, Kondoh M, Mitake T. Real-time Virtual Sonography for navigation during targeted prostate biopsy using magnetic resonance imaging data. Int J Urol. 2010 Oct;17(10):855-60. doi: 10.1111/j.1442-2042.2010.02612.x. Epub 2010 Aug 27. PMID 20807266
- [Background] Kuru TH, Roethke MC, Seidenader J, Simpfendorfer T, Boxler S, Alammar K, Rieker P, Popeneciu VI, Roth W, Pahernik S, Schlemmer HP, Hohenfellner M, Hadaschik BA. Critical evaluation of magnetic resonance imaging targeted, transrectal ultrasound guided transperineal fusion biopsy for detection of prostate cancer. J Urol. 2013 Oct;190(4):1380-6. doi: 10.1016/j.juro.2013.04.043. Epub 2013 Apr 19. PMID 23608676
- [Background] Chondros Kappa, Karpathakis Nu, Heretis Iota, Mavromanolakis Epsilon, Chondros N, Sofras F, Mamoulakis C. Validation of revised Epstein's criteria for insignificant prostate cancer prediction in a Greek subpopulation. Hippokratia. 2015 Jan-Mar;19(1):30-3. PMID 26435643
- [Background] Oon SF, Watson RW, O'Leary JJ, Fitzpatrick JM. Epstein criteria for insignificant prostate cancer. BJU Int. 2011 Aug;108(4):518-25. doi: 10.1111/j.1464-410X.2011.09979.x. Epub 2011 Feb 14. PMID 21320276
- [Background] Jeldres C, Suardi N, Walz J, Hutterer GC, Ahyai S, Lattouf JB, Haese A, Graefen M, Erbersdobler A, Heinzer H, Huland H, Karakiewicz PI. Validation of the contemporary epstein criteria for insignificant prostate cancer in European men. Eur Urol. 2008 Dec;54(6):1306-13. doi: 10.1016/j.eururo.2007.11.057. Epub 2007 Dec 7. PMID 18083294
- [Background] Sonn GA, Fan RE, Ghanouni P, Wang NN, Brooks JD, Loening AM, Daniel BL, To'o KJ, Thong AE, Leppert JT. Prostate Magnetic Resonance Imaging Interpretation Varies Substantially Across Radiologists. Eur Urol Focus. 2019 Jul;5(4):592-599. doi: 10.1016/j.euf.2017.11.010. Epub 2017 Dec 7. PMID 29226826
- [Background] Radtke JP, Wiesenfarth M, Kesch C, Freitag MT, Alt CD, Celik K, Distler F, Roth W, Wieczorek K, Stock C, Duensing S, Roethke MC, Teber D, Schlemmer HP, Hohenfellner M, Bonekamp D, Hadaschik BA. Combined Clinical Parameters and Multiparametric Magnetic Resonance Imaging for Advanced Risk Modeling of Prostate Cancer-Patient-tailored Risk Stratification Can Reduce Unnecessary Biopsies. Eur Urol. 2017 Dec;72(6):888-896. doi: 10.1016/j.eururo.2017.03.039. Epub 2017 Apr 8. PMID 28400169
- [Background] Roethke MC, Kuru TH, Mueller-Wolf MB, Agterhuis E, Edler C, Hohenfellner M, Schlemmer HP, Hadaschik BA. Evaluation of an Automated Analysis Tool for Prostate Cancer Prediction Using Multiparametric Magnetic Resonance Imaging. PLoS One. 2016 Jul 25;11(7):e0159803. doi: 10.1371/journal.pone.0159803. eCollection 2016. PMID 27454770